CLINICAL TRIAL: NCT00001959
Title: Pirfenidone in Focal Segmental Glomerulosclerosis:Phase II Study
Brief Title: Pirfenidone to Treat Kidney Disease (Focal Segmental Glomerulosclerosis)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jeffrey Kopp, M.D., Staff Clinician, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000042; 00-DK-0042
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Results first posted 2012-06-01 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2012-04

CONDITIONS: Fibrosis; Focal Glomerulosclerosis; Kidney Failure; Nephrotic Syndrome; Proteinuria
Keywords: Fibrosis; Nephrotic Syndrome; Proteinuria; Renal Failure; TGF-Beta; Focal Segmental Glomerulosclerosis; FSGS
MeSH Terms: conditions — Fibrosis; Glomerulosclerosis, Focal Segmental; Renal Insufficiency; Nephrotic Syndrome; Proteinuria; Camurati-Engelmann Syndrome | interventions — pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pirfenidone — During the study drug period of 12 months, patients will receive oral pirfenidone daily. For patients whose initial renal function is 50-80 ml/min as assessed by the MDRD equation, the initial pirfenidone dosage will be calculated at 40 mg/kg/d, with a maximum dose of 800 mg TID. For patients whose initial renal function is 30-50 ml/min, the initial dose will be 30 mg/kg/d. For patients whose initial renal function is between 15 and 30 ml/min, the initial dose will be 20 mg/kg/d.

SUMMARY:
This study will examine the effectiveness of the drug pirfenidone in treating focal segmental glomerulosclerosis (FSGS). Patients with this disease have kidney fibrosis (scarring) and proteinuria (excessive excretion of protein in the urine). About half of patients with FSGS eventually require kidney dialysis or transplant. Steroids, which are currently used to treat the disease, are effective in only a minority of patients. Other drugs, such as cyclosporin and cyclophosphamide, improve proteinuria in a very small percentage of patients and have serious side effects.

Patients with FSGS who wish to participate in this study will undergo pre-study evaluation with blood and urine tests. Patients must be on a stable dose of an ACE inhibitor (a drug that lowers blood pressure and reduces proteinuria) for at list 6 months before starting pirfenidone therapy. (Patients who are not already taking an ACE inhibitor will be started on the drug; those who cannot tolerate ACE inhibitors will be given a different drug.) Patients with elevated cholesterol will take a cholesterol-lowering drug. A diet containing approximately 1 gram of protein per kilogram of body weight per day will be recommended.

Patients will take pirfenidone by mouth 3 times a day for 12 months. Blood and urine will be tested once a month, either at NIH or by the patient's local kidney specialist. They will collect two 24-hour urine samples at the beginning of the treatment period, at 2-month intervals throughout the study, and at a 6-month follow-up. Patients will also be asked to give three to five tubes of blood and urine samples for analysis during the study.

In animal studies, pirfenidone improved kidney function and proteinuria and reduced kidney scarring in rats with a disease similar to FSGS. In human studies, pirfenidone improved breathing and survival in patients with lung fibrosis.

DETAILED DESCRIPTION:
The objective of this pilot phase II trial is to evaluate the ability of pirfenidone, a novel anti-fibrotic agent, to reduce the proteinuria and slow the rate of progression of renal insufficiency in patients with focal segmental glomerulosclerosis (FSGS). We will enroll 25 patients with renal biopsy proven FSGS and evidence of impaired renal function (glomerular filtration rate, GFR, of 10-80 ml/min; after 1/02 must have GFR greater than 25 ml/min) as assessed by the 4 variable Modification of Diet in Renal Disease equation. As standard of care therapy, all patients will also receive angiotensin converting enzyme inhibitor (ACEI) therapy, and will receive an HMG Co-A reductase inhibitor drug if hypercholesterolemic. Preliminary evaluation will assure that the patients meet the study requirements, and an evaluation period will be used to ensure that patients are on maximal conservative therapy prior to the baseline period. Patients will receive treatment with pirfenidone daily, with dose adjusted for body weight and level of kidney function. The primary end point will be the decrease glomerular filtration as a marker of glomerular injury; reduction in proteinuria will be a secondary end-point. If the pilot study suggests this drug delays progression of renal insufficiency or reduces proteinuria in patients with FSGS, we will proceed with a large scale randomized, placebo-controlled study.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adults greater than or equal to 18 years of age.
  2. Patients will provide informed consent.
  3. Biopsy proven FSGS.
  4. Glomerular filtration rate of at least 25 and no more than 80 ml/minute as assessed by the 4 variable Modification of diet in renal disease GFR equation.
  5. At least 6 months of renal function data must be available prior to the patient's receiving pirfenidone, and renal function must show a rate of decline of greater than or equal to 0.4 ml/min/month during this baseline period.
  6. Patients must have received no glucocorticoids, cyclophosphamide, mycophenolate or other immunosuppressive drugs for at least 2 months prior to the study period.
  7. Patients must have received no cyclosporin for at least 6 months prior to the study period.
  8. Patients must have been taking an angiotensin converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) at a stable dose for at least 6 months, unless intolerant of both classes of medication.
  9. Patients who are HIV seropositive will receive standard care for HIV disease (patients receiving immune-modulating therapy will be excluded).
  10. Women with child-bearing potential must maintain an effective birth control regimen (oral contraceptive, intrauterine device, barrier plus spermicide).
  11. Men will be advised that although Ames testing has been negative for any evidence of mutagenicity, they should consider use of contraceptives during the study period as well.

EXCLUSION CRITERIA:

1. Inability to give informed consent or cooperate with study.
2. Known intolerance to pirfenidone.
3. Evidence of FSGS associated with an additional primary or secondary glomerular disease (e.g. diabetes, membranous nephropathy, IgA nephropathy).
4. Recent (within 6 months) history of myocardial infarction.
5. History of peptic ulcer within 6 months.
6. History of cerebrovascular disease manifested by transient ischemic attack or cerebrovascular accident within 6 months.
7. Pregnancy, breast feeding or inadequate birth control.
8. History of photosensitivity dermatitis.
9. Concurrent drug treatment with gemfibrozil, cyclosporin or erythromycin, potassium-sparing diuretics and other drugs which may potentiate hyperkalemia, or concurrent immunosuppresive medications.
10. Requirement for NSAID therapy.
11. Requirement for interleukin-2 therapy or other immune-modulating medication.
12. Existence of any other condition which would complicate the implementation or interpretation of the study.
13. Renal transplant.
14. Evidence of significant hepatic disease, as indicated by serum transaminases greater than 3 times upper limit of normal, protime greater than 2 seconds prolonged.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 1999-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abbate M, Zoja C, Rottoli D, Corna D, Perico N, Bertani T, Remuzzi G. Antiproteinuric therapy while preventing the abnormal protein traffic in proximal tubule abrogates protein- and complement-dependent interstitial inflammation in experimental renal disease. J Am Soc Nephrol. 1999 Apr;10(4):804-13. doi: 10.1681/ASN.V104804. PMID 10203365
- [Background] Bodi I, Kimmel PL, Abraham AA, Svetkey LP, Klotman PE, Kopp JB. Renal TGF-beta in HIV-associated kidney diseases. Kidney Int. 1997 May;51(5):1568-77. doi: 10.1038/ki.1997.215. PMID 9150474
- [Background] Border WA, Noble NA. Transforming growth factor beta in tissue fibrosis. N Engl J Med. 1994 Nov 10;331(19):1286-92. doi: 10.1056/NEJM199411103311907. No abstract available. PMID 7935686
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2000-DK-0042.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 adults patients were enrolled between 2000-2004 at the clinical center of NIH
Period: Overall Study
Arm/Group | Pirfenidone
Started | 21
Completed | 18
Not Completed | 3
Not completed — newly diagnosed colon cancer | 1
Not completed — disabling sedation | 1
Not completed — non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pirfenidone
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
Baseline GFR [Mean (Standard Deviation); unit: ml/min/1.73 m^2] | 26.0 (9.4)
Baseline period proteinuria [Median (Inter-Quartile Range); unit: g/d] | 3.2 [1.6 to 4.4]
Decrease in GFR during baseline period [Median (Inter-Quartile Range); unit: ml/min/1.73 m^2] | -0.61 [-1.31 to -0.41]
Duration of angiotensin antagonist therapy before treatment [Median (Inter-Quartile Range); unit: month] — 2 patients did not receive angiotensin antagonist therapy during the baseline periods because of angioedema and hypotension.
  month | 15 [8.4 to 33]

OUTCOME MEASURES:

1. Primary Outcome: Decrease in GFR During Treatment Period
Time Frame: 12 months from baseline
Population: ITT
Measure: Mean (Inter-Quartile Range); unit: ml/min/1.73 m2
Arm/Group | Pirfenidone
Number analyzed (Participants) | 18
ml/min/1.73 m2 | -0.45 [-0.78 to -0.16]
Statistical Analysis 1: Comparison: Pirfenidone; H0: GFR Decrease during baseline period and treatment period are same; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Proteinuria After Treatment
Time Frame: 12 months from baseline
Measure: Median (Inter-Quartile Range); unit: g/d
Arm/Group | Pirfenidone
Number analyzed (Participants) | 18
g/d | 4.3 [1.2 to 6.7]
Statistical Analysis 1: Comparison: Pirfenidone; H0: Proteinuria during baseline and treatment periods are same; Test type: Superiority or Other; p = 0.16, Kruskal-Wallis

3. Secondary Outcome: Proportion of Patients With Positive Change in GFR
Time Frame: 12 months from baseline
Measure: Number; unit: participants
Arm/Group | Pirfenidone
Number analyzed (Participants) | 18
participants | 13

ADVERSE EVENTS:
Time Frame: 60 months
Description: Include all adverse events either judged to be related to the study or unrelated to the study
Arm/Group | Pirfenidone
Serious Adverse Events (participants affected / at risk) | 3/21
Other Adverse Events (participants affected / at risk) | 16/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pirfenidone (N=21)
Death (unrelated to the trial) (Injury, poisoning and procedural complications) | 1 (1) — traumatic subdural hematoma
Colon cancer (unrelated to the trial) (Gastrointestinal disorders) | 1 (1)
elevated liver enzymes (judged possibly related to the trial) (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pirfenidone (N=21)
Gastrointestinal discomfort (Gastrointestinal disorders) | 8 (8)
Sedation or fatigue (General disorders) | 6 (6)
photosensitivity dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
No control group, measurement imprecision, results may not applicable to all patients with FSGS, needs histologic evidence to support our findings, Optimal dosage needs to be identified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes